CLINICAL TRIAL: NCT07109752
Title: Effect of Mindfulness-based eHealth Cardiac Rehabilitation on Psychological Wellbeing and Risk Factor Management of Patients With Coronary Heart Disease: A Randomized Controlled Trial
Brief Title: Effect of eHealth Cardiac Rehabilitation Incorporating Mindfulness for Patients With Coronary Heart Disease
Acronym: eCR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tung Wah College (Other)
Responsible Party: Principal Investigator, SU JingJing, Assistant Professor, Tung Wah College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TungWC REC2024214; REC2024214 (Other: Tung Wah College)
Record Dates: First submitted 2025-07-18; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Coronary Heart Disease (CHD)
Keywords: cardiac rehabilitation; mindfulness; eHealth
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eCR (Experimental): Intervention arm
  Interventions: Behavioral: eHealth cardiac rehabilitation
- Control (No Intervention): Usual care

INTERVENTIONS:
Behavioral: eHealth cardiac rehabilitation — A face-to-face interview for goal setting and action planning, as well as learning the use of CR website and accelerometer.
  Arms: eCR

SUMMARY:
People with coronary heart disease (CHD) often feel more stressed, which can increase the risk of having another heart problem. Cardiac rehabilitation (CR) is a common treatment for those with CHD, focusing on changing lifestyles and managing the disease. However, it often does not address stress management adequately. There is also a lack of psychological therapy and involvement of mental health professionals in online CR programs. Because traditional CR programs have low participation rates, online platforms are becoming more popular for providing rehabilitation support. This is important because more than half of people with CHD report high stress levels, which can cause or worsen heart problems. To address this issue, the proposed study will test an online CR program that includes mindfulness to help manage stress for CHD patients.

DETAILED DESCRIPTION:
The proposed project is a study designed to test the effects of an online cardiac rehabilitation program, which includes mindfulness, on stress and health outcomes for people with coronary heart disease (CHD). The study will last 12 weeks and will be structured as a single-blinded, two-group randomized controlled trial. This means that participants will be randomly assigned to either the treatment group or a control group, and they won't know which group they're in. After the trial, there will be an evaluation to gather more in-depth insights.

Participants will be asked to complete assessments using questionnaires and activity monitors at the start of the study, at 6 weeks, and at 12 weeks. Each assessment will take about 40 minutes, and there will also be a 30 to 40-minute interview.

Those in the intervention group will have a face-to-face meeting to set goals and learn how to use the CR website and activity monitors, which will take about 50 minutes. They will be encouraged to use the website weekly to learn about healthy lifestyle changes, like walking briskly for 30 minutes a day, eating a healthy diet, listening to mindfulness audios, and not smoking. A nurse will call them every two weeks for the first six weeks to check in.

The study is led by an Assistant Professor who has the necessary office space and access to various facilities to support the research. She specializes in cardiovascular health and has established connections in the field of cardiac rehabilitation, which are valuable for successfully conducting the study.

The team includes co-investigators with expertise in physiotherapy, exercise rehabilitation, psychiatric nursing, and intensive care nursing, ensuring the study is well-supported and that results are properly reported and published.

ELIGIBILITY:
Inclusion Criteria:

People will be eligible for this study if they were:

1. diagnosed with CHD (within the past 6 months),
2. undergone conservative treatment, such as percutaneous coronary intervention (PCI) and/ or medication,
3. currently under stable medication regimen and discharged to home.
4. aged 18 years or older,
5. reported scores ranging from 3 (to some degree) to 5 (very much) scores on a single-item stress symptoms scale (Elo et al., 2003),
6. using a computer and/or smartphone to access the Internet at home,
7. and, read and speak Chinese.

Exclusion Criteria:

1. diagnosis of acute psychotic disease;
2. presence of a life-limiting condition;
3. prescribed contradictions to physical activity; and,
4. presence of hearing, visual, or ambulatory disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2024-07-20 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Perceived stress level | baseline, 6-week, 12- week
  The Perceived Stress Scale (PSS-10), with total scores ranging from 0 to 40 and higher scores indicating higher psychological stress

SECONDARY OUTCOMES:
Anxiety level | baseline, 6-week, 12-week
  Generalized Anxiety Disorder 7-item, seven items ranges from 0 to 21 scores. 0-4: minimal anxiety. 5-9: mild anxiety. 10-14: moderate anxiety. 15-21: severe anxiety.
Depression level | baseline, 6-week, 12-week
  Patient Health Questionnaire (PHQ-9) with total scores of 5, 10, 15, and 20 represent cutpoints for mild, moderate, moderately severe and severe depression, respectively.
Physical activity | baseline, 6-week, 12-week
  Daily steps measured by accelerometer
Sleep | baseline, 6-week, 12-week
  Sleep time measured by accelerometer
Health Related Quality of life | baseline, 6-week, 12-week
  Short-Form Six Dimensions (SF-6D), six items ranged from 6- 37 scores, with higher score indicate lower quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Tung Wah College, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Participants may not have given explicit consent for their data to be shared beyond the initial study, limiting the ability to share their data legally and ethically.

REFERENCES:
- [Background] Batalik L, Filakova K, Sladeckova M, Dosbaba F, Su J, Pepera G. The cost-effectiveness of exercise-based cardiac telerehabilitation intervention: a systematic review. Eur J Phys Rehabil Med. 2023 Apr;59(2):248-258. doi: 10.23736/S1973-9087.23.07773-0. Epub 2023 Jan 24. PMID 36692413

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-17): https://cdn.clinicaltrials.gov/large-docs/52/NCT07109752/Prot_SAP_000.pdf